CLINICAL TRIAL: NCT02989649
Title: A Prospective, Non-Interventional Study of the Use of Alogliptin and Alogliptin Fixed-Dose Combinations With Pioglitazone and With Metformin in Standard Clinical Practice
Brief Title: Non-Interventional Study of the Use of Alogliptin and Alogliptin Fixed-Dose Combinations With Pioglitazone and With Metformin in Standard Clinical Practice
Status: Terminated | Type: Observational
Why Stopped: Business Decision; No Safety Or Efficacy Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Alogliptin-5009
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Pioglitazone; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alogliptin or Alogliptin Fixed Dose Combinations (FDCs): Participants with type 2 diabetes mellitus (T2DM) who received alogliptin or alogliptin FDCs, orally, prescribed by the physician as part of participants' T2DM treatment program (independent of participation in this study) were observed for approximately 6 months, or up to loss to follow-up or death, whichever occurred first.
  Interventions: Drug: Alogliptin; Drug: Alogliptin FDC With Pioglitazone; Drug: Alogliptin FDC With Metformin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
Drug: Alogliptin FDC With Pioglitazone — Alogliptin FDC with pioglitazone tablets
Drug: Alogliptin FDC With Metformin — Alogliptin FDC with metformin tablets

SUMMARY:
The purpose of this study is to observe alogliptin and alogliptin fixed-dose combinations (FDCs) utilization patterns, as well as clinical response to treatment with alogliptin or alogliptin FDCs, in standard clinical practice.

DETAILED DESCRIPTION:
The drug being studied in this study is called alogliptin and alogliptin FDCs. Alogliptin and alogliptin FDCs is being researched to treat people who have diabetes mellitus type 2. This study will look at the glycosylated hemoglobin (HbA1c) level dynamics in participants with diabetes mellitus type 2.

The study enrolled 593 patients. Alogliptin and alogliptin FDCs will be prescribed by the physician as part of participants' T2DM treatment program (independent of participation in this study).

This multi-center study will be conducted in China. The overall duration of study for observation will be approximately 6 months, or up to loss to follow-up or death, whichever occurs first. Participants will make multiple visits to the clinic as per regular doctor's appointments.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of T2DM.
2. Has made the decision, along with his/her treating physician, to begin treatment with alogliptin or alogliptin fixed-dose combinations (FDCs).
3. Has an glycated hemoglobin (HbA1c) value recorded at most 3 months before initiation of treatment with alogliptin or alogliptin FDCs.
4. Alogliptin or alogliptin FDCs is prescribed according to the approved label for China and Hong Kong.

Exclusion Criteria:

1. Has gestational diabetes or type 1 diabetes mellitus.
2. Has used Dipeptidyl peptidase-4 inhibitors (DPP-IV inhibitors) or Glucagon like peptide-1 agonists (aGLP-1) within the 3 months prior to the start of alogliptin or alogliptin FDCs treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with type 2 diabetes mellitus (T2DM) will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 593 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (11):
- China (9):
  - Beijing, Beijing Municipality
  - Wuhan, Hubei
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - Jinan, Shandong
  - Qingdao, Shandong
  - Taian, Shandong
  - Tai’an, Shandong
  - Tianjin, Tianjin Municipality
- Hong Kong (2):
  - Sai Ying Pun
  - Shatin

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in China from 22 Dec 2016 to 26 Jan 2018.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus (T2DM) prescribed alogliptin or alogliptin Fixed Dose Combinations (FDCs) with either metformin or pioglitazone were enrolled in this observational study.
Period: Overall Study
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Started | 593
Started But Not Treated | 84
Eligible to Enter Into Treatment Period | 509
Completed | 173
Not Completed | 420
Not completed — Patient/Investigator's Decision to Stop | 403
Not completed — Adverse Event/Adverse Drug Reaction | 1
Not completed — Lost For Observation During Study | 3
Not completed — Reason Not Specified | 13

BASELINE CHARACTERISTICS:
Population: All participants dosed included participants with complete demographic information and eligible for the study and dosed at least once.
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.65)
Age, Customized [Count of Participants; unit: Participants]
  <45 years | 92
  >=45 to <65 years | 309
  >=65 years | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207
  Male | 302
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 508
  White | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Nationality | 504
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  China | 509
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with evaluable data for this baseline measure.
  cm
    number analyzed (Participants) | 500
    (all) | 167.37 (8.089)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with evaluable data for this baseline measure.
  kg
    number analyzed (Participants) | 500
    (all) | 72.66 (12.208)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index(BMI)=weight (kg)/[height (m)^2]. BMI is calculated using the participant's baseline height and weight measurement. Population: Number analyzed is the number of participants with evaluable data for this baseline measure.
  kg/m^2
    number analyzed (Participants) | 500
    (all) | 25.86 (3.500)
Body Mass Index, Customized [Count of Participants; unit: Participants] — Body Mass Index(BMI)=weight (kg)/[height (m)^2]. BMI is calculated using the participant's baseline height and weight measurement.
  Participants
    <25 kg/m^2 | 193
    25 to <30 kg/m^2 | 256
    >=30 kg/m^2 | 51
    Missing | 9
Glycosylated hemoglobin (HbA1c) Level [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Glycosylated hemoglobin is the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound. Glycosylated hemoglobin as a diagnostic criteria of diabetes mellitus is ≥6.5%. Population: Number analyzed is the number of participants with evaluable data for this baseline measure.
  percentage of glycosylated hemoglobin
    number analyzed (Participants) | 498
    (all) | 8.690 (1.8807)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Level at Month 6
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Glycosylated hemoglobin (HbA1c) as a diagnostic criteria of diabetes mellitus is ≥6.5%. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 6
Population: All participants dosed included participants with complete demographic information and eligible for the study and dosed at least once. Overall number of participants analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 140
percentage of glycosylated hemoglobin | -1.092 (1.6803)
Statistical Analysis 1: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for data at Baseline compared to the data at Month 6; Test type: Other; p < 0.001, Regression, Linear; Least Square Mean (LSM) = -1.25, 95% CI 2-sided [-1.44 to -1.05], Standard Error of Mean 0.098 — The LSM and CI are from Mixed effect Model Repeat Measurement (MMRM) model, that used visit as a predictor and baseline value as a covariate. For change from baseline, covariance structure=Unstructured

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Level at Month 6 in Subgroups of Participants With Different Clinical Characteristics
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Month 6 relative to baseline. Glycosylated hemoglobin (HbA1c) as a diagnostic criteria of diabetes mellitus is ≥6.5%. Subgroups included participants with different baseline clinical characteristics with predictors such as prior therapy of diabetes mellitus, sex, age group, cardiovascular risk group, therapy type (monotherapy or combined therapy), baseline body mass index (BMI) and initial glycemic control. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 140
percentage of glycosylated hemoglobin
  Prior Therapy of Diabetes Mellitus, Ever Used: number analyzed (Participants) | 108
  Prior Therapy of Diabetes Mellitus, Ever Used | -1.154 (1.7555)
  Prior Therapy of Diabetes Mellitus, Never Used: number analyzed (Participants) | 32
  Prior Therapy of Diabetes Mellitus, Never Used | -0.882 (1.4015)
  Sex, Male: number analyzed (Participants) | 86
  Sex, Male | -1.055 (1.5898)
  Sex, Female: number analyzed (Participants) | 54
  Sex, Female | -1.150 (1.8292)
  Age, <45 years: number analyzed (Participants) | 23
  Age, <45 years | -1.658 (1.8206)
  Age, >=45 to <65 years: number analyzed (Participants) | 78
  Age, >=45 to <65 years | -1.370 (1.7121)
  Age,>=65 years: number analyzed (Participants) | 39
  Age,>=65 years | -0.203 (1.1423)
  Cardiovascular Risk Group, Yes: number analyzed (Participants) | 7
  Cardiovascular Risk Group, Yes | -1.100 (2.4973)
  Cardiovascular Risk Group, No: number analyzed (Participants) | 133
  Cardiovascular Risk Group, No | -1.092 (1.6400)
  Therapy Type, Monotherapy: number analyzed (Participants) | 26
  Therapy Type, Monotherapy | -1.032 (1.5122)
  Therapy Type, Combined Therapy: number analyzed (Participants) | 114
  Therapy Type, Combined Therapy | -1.106 (1.7222)
  Baseline BMI, <25 kg/m^2: number analyzed (Participants) | 64
  Baseline BMI, <25 kg/m^2 | -1.101 (1.7339)
  Baseline BMI, 25 to <30 kg/m^2: number analyzed (Participants) | 64
  Baseline BMI, 25 to <30 kg/m^2 | -1.037 (1.6151)
  Baseline BMI, >=30 kg/m^2: number analyzed (Participants) | 12
  Baseline BMI, >=30 kg/m^2 | -1.342 (1.8530)
  Initial Glycemic Control, <7%: number analyzed (Participants) | 41
  Initial Glycemic Control, <7% | -0.046 (0.7345)
  Initial Glycemic Control, >=7%: number analyzed (Participants) | 99
  Initial Glycemic Control, >=7% | -1.525 (1.7713)
Statistical Analysis 1: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Prior therapy of diabetes mellitus, Ever used or Never used; Test type: Other; p = 0.423, Regression, Linear
Statistical Analysis 2: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Sex, Male or Female; Test type: Other; p = 0.747, Regression, Linear
Statistical Analysis 3: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Age, <45 or >=45 to <65 years or >=65 years; Test type: Other; p < 0.001, Regression, Linear
Statistical Analysis 4: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Cardiovascular risk group, Yes or No; Test type: Other; p = 0.990, Regression, Linear
Statistical Analysis 5: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Therapy type, Monotherapy or Combined therapy; Test type: Other; p = 0.841, Regression, Linear
Statistical Analysis 6: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Baseline BMI, <25 or 25 to <30 or >=30 kg/m^2; Test type: Other; p = 0.847, Regression, Linear
Statistical Analysis 7: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for subgroup: Initial glycemic control, <7% or >=7%; Test type: Other; p < 0.001, Regression, Linear

3. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c Level by <7.0%
Description: Percentage of participants with a decrease of <7.0% from baseline in HbA1c were reported.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 147
percentage of participants | 51.0 [0.43 to 0.59]

4. Secondary Outcome: Percentage of Participants With a Decrease in HbA1c Level by >0.3% and No Tolerability Findings
Description: Percentage of participants with a decrease of >0.3% from baseline in HbA1c along with no tolerability findings were reported. Tolerability findings included hypoglycemic event, or weight gain ≥5%.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 140
percentage of participants | 64.3 [0.56 to 0.72]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) Level Over Time
Description: The change between the fasting plasma glucose value collected at Months 3 and 6 relative to baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3 and 6
Population: All participants dosed included participants with complete demographic information and eligible for the study and dosed at least once. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 509
mg/dL
  Month 3: number analyzed (Participants) | 213
  Month 3 | -1.058 (3.0026)
  Month 6: number analyzed (Participants) | 82
  Month 6 | -0.714 (2.9802)
Statistical Analysis 1: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for data at Baseline compared to the data at Month 3; Test type: Other; Least Square Mean (LSM) = -0.95, 95% CI 2-sided [-1.29 to -0.62], Standard Error of Mean 0.170 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for data at Baseline compared to the data at Month 6; Test type: Other; Least Square Mean (LSM) = -0.87, 95% CI 2-sided [-1.36 to -0.39], Standard Error of Mean 0.245 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) Level Over Time
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Months 3 and 6 relative to baseline. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Months 3 and 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 509
percentage of glycosylated hemoglobin
  Month 3: number analyzed (Participants) | 332
  Month 3 | -1.022 (2.3669)
  Month 6: number analyzed (Participants) | 140
  Month 6 | -1.092 (1.6803)
Statistical Analysis 1: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for data at Baseline compared to the data at Month 3; Test type: Other; Least Square Mean (LSM) = -0.95, 95% CI 2-sided [-1.18 to -0.72], Standard Error of Mean 0.117 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Alogliptin or Alogliptin Fixed Dose Combinations (FDCs); Statistical analysis for data at Baseline compared to the data at Month 6; Test type: Other; Least Square Mean = -1.25, 95% CI 2-sided [-1.44 to -1.05], Standard Error of Mean 0.098 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An ADR is defined as any response to a medicinal product that is noxious and unintended and that occurs at doses normally used in humans for the prophylaxis, diagnosis, or therapy of diseases or for the restoration, correction, or modification of physiological function. An SAE is defined as any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically important due to other reasons than the above mentioned criteria. Adverse events such as pancreatitis, hepatic disorders, and hypersensitivity reactions (including angioedema, anaphylaxis, and Stevens-Johnson syndrome) were considered as AESI.
Time Frame: Baseline up to Month 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 509
Participants
  Adverse Drug Reaction (ADR) | 1
  Serious Adverse Event (SAE) | 0
  Adverse Event of Special Interest (AESI) | 0

8. Secondary Outcome: Percentage of Participants Who Remain on Treatment With Alogliptin or Alogliptin FDCs
Time Frame: Months 3 and 6
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 509
percentage of participants
  Month 3: number analyzed (Participants) | 380
  Month 3 | 100
  Month 6: number analyzed (Participants) | 154
  Month 6 | 100

9. Secondary Outcome: Time to Alogliptin or Alogliptin FDCs Dose Escalation or Dose Reduction
Time Frame: Months 3 and 6
Population: No participant was experienced the dose adjustment (dose escalation or dose reduction).
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Month 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs)
All-Cause Mortality (participants affected / at risk) | 0/509
Serious Adverse Events (participants affected / at risk) | 0/509
Other Adverse Events (participants affected / at risk) | 55/509
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin or Alogliptin Fixed Dose Combinations (FDCs) (N=509)
Abdominal discomfort (Gastrointestinal disorders) | 48
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Hypertension (Vascular disorders) | 2
Gastroenteritis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02989649/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT02989649/SAP_001.pdf